CLINICAL TRIAL: NCT03784586
Title: The Electrophysiological Study Guided ICD Strategy in Prevention of Arrhythmic Cardiac Death in Myotonic Dystrophy Type 1 Patients With Conduction System Disease (ACADEMY 1 Study)
Brief Title: Sudden Cardiac Death Stratification in Myotonic Dystrophy Type 1 Patients
Acronym: ACADEMY 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Vincenzo Russo, MD, PhD, Assistant Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 01_MD1
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Myotonic Dystrophy 1; Sudden Cardiac Death
Keywords: Arrhythmias; electrophisiological study; primary prevention
MeSH Terms: conditions — Myotonic Dystrophy; Death, Sudden, Cardiac; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive EPS - ICD: Patients with inducible sustained ventricular tachycardia or ventricular fibrillation at EPS evaluation underwent ICD implantation
- Negative EPS - PMK: All non inducible patients underwent PMK implantation

SUMMARY:
The aim of the study is to evaluate if the electrophysiological study (EPS) guided therapy, including the prophylactic implantation of implantable cardioverter defibrillator (ICD), in inducible patients, is able to improve survival in comparison with conventional therapy (CONV strategy) in Myotonic Dystrophy type 1 patients with conduction disorders.

DETAILED DESCRIPTION:
Trial design:

This is a double-arm prospective observational study.

Patient population:

To be included in the study, DM1 patients had to have at least 18 years old, LVEF >35% on two-dimensional echocardiography, permanent pacing indication after non-invasive electrocardiographic evaluation or invasive EPS evaluation, according to the current guidelines. The following exclusion criteria were applied: electrolyte imbalance, thyroid disorders, prior cardiac surgery, prior cardiac arrest, prior spontaneous sustained ventricular arrhythmias, absuntion of antiarrhythmic drugs or medication known to affect cardiac conduction. All eligible DM1 patients underwent EPS for programmed ventricular stimulation; those in whom a sustained ventricula arrhythmia was inducible underwent subsequently ICD implantation. Non-inducible DM1 patients did not receive an ICD and underwent pacemaker implantation.

Endpoints:

The primary endpoint was all-cause mortality. Secondary end-points were sudden death (SD), death due to cardiac arrhythmias, ICD interventions and arrhythmic events in implanted patients.

ELIGIBILITY:
Inclusion Criteria:

* MD1 diagnosis genetically confirmed
* LVEF >35% on two-dimensional echocardiography
* Permanent pacing indication according to the current guidelines

Exclusion Criteria:

* Electrolyte imbalance
* Thyroid disorders
* Prior cardiac surgery
* Prior cardiac arrest
* Prior spontaneous sustained ventricular arrhythmias

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD1 patients with permanent pacing indication and needed of sudden cardiac death screening.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Sudden Cardiac Death | 24 months

SECONDARY OUTCOMES:
All-cause mortality | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vincenzo Russo, Naples, Italy

IPD SHARING:
Plan to Share IPD: No